CLINICAL TRIAL: NCT04207333
Title: The Combined Effects of Prolonged Sitting and Mental Stress on Vascular and Cerebrovascular Function in Middle-Aged Adults
Brief Title: Combined Effects of Prolonged Sitting and Mental Stress on the Cardiovascular System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19-1843; 2KR1211907 (Other Grant/Funding Number: NCTraCS)
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2020-03

CONDITIONS: Sedentary Behavior; Cardiovascular Risk Factor; Mental Stress; Cognitive Change; Cerebrovascular Insufficiency
MeSH Terms: conditions — Sedentary Behavior; Stress, Psychological; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be exposed to mental stress following either 20 min or 120 min sitting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Sitting + Mental Stress, Then Brief Sitting + Mental Stress (Experimental): Participants will sit for 120 min prior to being exposed to mental stress Following 10 minutes of supine rest, participants will switch to an upright sitting position and remain seated for 120 minutes while watching a documentary. Following the 10 minutes quiet rest the participants will be subjected to a 5 minute mental arithmetic test. Following a 2-5 day wash-out period, participants will be exposed to the other condition (brief sitting, followed by mental stress). For this condition participants will rest in the supine position for 10 minutes, then will be switched to an upright seated position. Following the 10 minutes quiet rest in the seated position, participants will be subjected to a 5 minute mental arithmetic test.
  Interventions: Behavioral: Mental Arithmetic Test
- Brief Sitting + Mental Stress, Then Prolonged Sitting + Mental Stress (Experimental): Following 10 minutes of supine rest, participants will switch to an upright sitting position and remain seated for 10 minutes. Following the 10 minutes quiet rest the participants will be subjected to a 5 minute mental arithmetic test. Following a 2-5 day wash-out period, participants will be exposed to the other condition (prolonged sitting, followed by mental stress). For this condition participants will rest in the supine position for 10 minutes, then will be switched to an upright seated position. Participants will sit quietly for 120 min while watching a documentary, following which the participants will be subjected to a 5 minute mental arithmetic test.
  Interventions: Behavioral: Mental Arithmetic Test

INTERVENTIONS:
Behavioral: Mental Arithmetic Test — The researcher will call out a four-digit number and ask the participant to subtract either 7 or 13. Each minute, a new four-digit number will be called out and the participant must subtract the 7 or 13 from the number. The test will last approximately 5 minutes
  Other Names: Mental Stressor

SUMMARY:
Prolonged sitting may pose a public health risk through its effects on the cardiovascular system, and may lead to impaired whole-body cardiovascular health, which includes both vascular and cerebrovascular function. These effects may interact with other environmental variables, such as stress. However, no study has investigated the combined effect of a mental stressor and prolonged sitting on vascular and cerebrovascular function. The combined effect of prolonged sitting and mental stress may lead to an exacerbated effect on vascular, cerebrovascular, and executive function. The investigators hypothesize that mental stress with the addition of prolonged sitting [PS] will result in a greater increase in peripheral, central and cerebral arterial stiffness and elicit a decrease in cerebral perfusion, total blood flow to the brain, middle cerebral artery velocity and executive function, compared to mental stress without prolonged sitting [CON]. The findings from this study may result in a public health message regarding sedentary behavior and stress, and will help elucidate the mechanisms behind acute vascular, cerebrovascular, and cognitive dysfunction during prolonged sitting.

DETAILED DESCRIPTION:
This study is a multi-visit (three in total) randomized crossover trial. During a single familiarization session, the research team will obtain informed consent, and will describe to participants the purposes and procedures of this study. They will then be exposed to all experimental devices on in a quiet, dimly lit and environmentally controlled room. Participants will return to the same location for two experimental conditions following these pre-assessment guidelines:

* Fasted (> 12 hours), consuming only water.
* No caffeine consumption 12 hours prior to testing.
* No vigorous exercise 24 hours prior to testing.
* No alcohol consumption 24 hours prior to testing.

Participants will arrive to the Applied Physiology Laboratory between 6:00 and 10:00 a.m. fasted (for Visit 3: 2-5 days following the Visit 2). Participants will be fasted and refrain from caffeine intake for at least 12 hours, and alcohol and strenuous physical activity for at least 24 hours prior to arrival. Upon arrival, height and weight will be recorded followed by 10 minutes of quiet rest in the supine position. During these 10 minutes, the subject will be fitted with a Near Infra-Red Spectroscopy probe on the prefrontal cortex and medial gastrocnemius. The non-invasive continuous blood pressure, transcranial doppler, and Vicorder arterial stiffness devices will also be affixed to the participant during this time period during this time. Sitting periods will begin for both conditions once all devices are attached to the participant, the subject is shifted to an upright seated position, and at least 10 minutes of supine rest has been recorded. During the control (CON) visit, subjects will undergo a brief 20 minute sitting period. For the prolonged sitting (PS) condition, subjects will be asked to sit still and quietly for 2 hours while watching a non-stimulating documentary. Each condition will receive the mental stress at the conclusion of the sitting periods in both CON and PS. After exposure to the mental stress in both conditions, data collection procedures for this protocol will be completed. Arterial stiffness measurements will be made immediately after the mental stress, and then every 5 minutes, up to 30 minutes. Brain blood flow will be assessed by ultrasound after completion of the arterial stiffness measures. Finally, a battery of cognitive tests (Verbal Fluency Test and Trails A+B tests) will be administered to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female

Exclusion Criteria:

* Any known cardio-metabolic disorders
* Taking medications known to affect cardiovascular function
* Report drug or alcohol abuse
* Report cigarette smoking
* Pregnant women

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jade Blackwell, MS, Principal Investigator — University of North Carolina, Chapel Hill; Lee Stoner, PhD, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: One year after study completion.
Access Criteria: After the results of the research questions outlined in the grant are published, the investigators will share the study protocol, statistical analysis plan, analytical plan, and deidentified data. Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Prolonged Sitting + Mental Stress, Then Brief Sitting + Mental Stress: Participants will sit for 120 min prior to being exposed to mental stress Following 10 minutes of supine rest, participants will switch to an upright sitting position and remain seated for 120 minutes while watching a documentary. Following the 10 minutes quiet rest the participants will be subjected to a 5 minute mental arithmetic test. Following a 2-7 day wash-out period, participants will be exposed to the other condition (brief sitting, followed by mental stress). For this condition participants will rest in the supine position for 10 minutes, then will be switched to an upright seated position. Following the 10 minutes quiet rest in the seated position, participants will be subjected to a 5 minute mental arithmetic test.
  Mental Arithmetic Test: The researcher will call out a four-digit number and ask the participant to subtract either 7 or 13. Each minute, a new four-digit number will be called out and the participant must subtract the 7 or 13 from the number. The test will last approximately 5 minutes
- Brief Sitting + Mental Stress, Then Prolonged Sitting + Mental Stress: Following 10 minutes of supine rest, participants will switch to an upright sitting position and remain seated for 10 minutes. Following the 10 minutes quiet rest the participants will be subjected to a 5 minute mental arithmetic test. Following a 2-7 day wash-out period, participants will be exposed to the other condition (prolonged sitting, followed by mental stress). For this condition participants will rest in the supine position for 10 minutes, then will be switched to an upright seated position. Participants will sit quietly for 120 min while watching a documentary, following which the participants will be subjected to a 5 minute mental arithmetic test.
  Mental Arithmetic Test: The researcher will call out a four-digit number and ask the participant to subtract either 7 or 13. Each minute, a new four-digit number will be called out and the participant must subtract the 7 or 13 from the number. The test will last approximately 5 minutes
Period: First Intervention (Single 1-Day Visit)
Arm/Group | Prolonged Sitting + Mental Stress, Then Brief Sitting + Mental Stress | Brief Sitting + Mental Stress, Then Prolonged Sitting + Mental Stress
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Washout (2-7 Days)
Arm/Group | Prolonged Sitting + Mental Stress, Then Brief Sitting + Mental Stress | Brief Sitting + Mental Stress, Then Prolonged Sitting + Mental Stress
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Second Intervention (Single 1-Day Visit)
Arm/Group | Prolonged Sitting + Mental Stress, Then Brief Sitting + Mental Stress | Brief Sitting + Mental Stress, Then Prolonged Sitting + Mental Stress
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who completed both conditions in either Period 1 or Period 2 or Period 3 as per randomization schedule.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Brachial-femoral Pulse Wave Velocity (bfPWV)
Description: bfPWV (m/s) is the velocity at which a pressure wave travels between the brachial and femoral arterial segments. An increase in bfPWV represents increased arterial stiffness (worse outcome).
Time Frame: Baseline and immediately following the acute mental stressor
Measure: Mean (Standard Error); unit: m/s
Groups:
- Prolonged Sitting With Mental Stress: Participants will sit for 120 min prior to being exposed to mental stress Following 10 minutes of supine rest, participants will switch to an upright sitting position and remain seated for 120 minutes while watching a documentary. Following the 10 minutes quiet rest the participants will be subjected to a 5 minute mental arithmetic test.
  Mental Arithmetic Test: The researcher will call out a four-digit number and ask the participant to subtract either 7 or 13. Each minute, a new four-digit number will be called out and the participant must subtract the 7 or 13 from the number. The test will last approximately 5 minutes
- Brief Sitting With Mental Stress: Following 10 minutes of supine rest, participants will switch to an upright sitting position and remain seated for 10 minutes. Following the 10 minutes quiet rest the participants will be subjected to a 5 minute mental arithmetic test.
  Mental Arithmetic Test: The researcher will call out a four-digit number and ask the participant to subtract either 7 or 13. Each minute, a new four-digit number will be called out and the participant must subtract the 7 or 13 from the number. The test will last approximately 5 minutes
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 6 | 6
m/s | -0.26 (0.56) | 0.22 (0.56)

2. Primary Outcome: Change in Heart-middle Cerebral Artery Pulse Wave Velocity (Brain PWV)
Description: Brain PWV (cm/s) is the velocity at which a pressure wave travels between the heart and cerebrovascular system. An increase in Brain PWV represents increased arterial stiffness (worse outcome).
Time Frame: Baseline and immediately following the acute mental stressor
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 6 | 6
cm/s | 6.1 (2.8) | -0.97 (2.8)

3. Secondary Outcome: Mean Change Carotid-femoral Pulse Wave Velocity (PWV)
Description: Carotid PWV (m/s) is the velocity at which a pressure wave travels between the carotid and femoral arterial segments. An increase in carotid PWV represents increased arterial stiffness (worse outcome).
Time Frame: Baseline and immediately following the acute mental stressor
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 6 | 6
m/s | -0.26 (0.56) | 0.22 (0.56)

4. Secondary Outcome: Mean Change in Femoral-ankle PWV
Description: Femoral-ankle PWV (m/s) is the velocity at which a pressure wave travels between the femoral-ankle arterial segments. An increase in femoral-ankle PWV represents increased arterial stiffness (worse outcome).
Time Frame: Baseline and immediately following the acute mental stressor
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 6 | 6
m/s | 1.28 (1.00) | 1.20 (1.00)

5. Secondary Outcome: Mean Change Augmentation Index
Description: Augmentation Index is a measure of arterial wave reflection and calculated as augmentation pressure divided by central pulse pressure.
Time Frame: Baseline and immediately following the acute mental stressor
Measure: Mean (Standard Error); unit: percentage of pulse pressure
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 6 | 6
percentage of pulse pressure | -1.83 (4.25) | -1.92 (4.25)

6. Secondary Outcome: Mean Executive Function
Description: Executive Function was measured at the end of each condition by recording the completion time of a trail making test. The trail making test was delivered using a tablet and the time to complete the test was recorded. Subject instructed to connect a set of 25 dots as rapidly as possible.
Time Frame: following the acute mental stressor
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 6 | 6
sec | 48.7 (20.2) | 76.2 (75.2)

7. Secondary Outcome: Neurovascular Coupling
Description: Neurovascular Coupling reflects the cerebral blood flow during a cognitive task.
Time Frame: following the acute mental stressor
Population: This data was not collected.
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the intervention up to a total of approximately 8 days
Arm/Group | Prolonged Sitting With Mental Stress | Brief Sitting With Mental Stress
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT04207333/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT04207333/ICF_001.pdf